CLINICAL TRIAL: NCT04173910
Title: Effect of the Left Paratracheal Compression of the Cervical Esophagus and the Sellick Manoeuvre on the Compressibility of the Carotid Artery and Its Possible Effects on the Vascular Flow
Brief Title: Carotid Artery Analysis During an LPEC Manoeuvre
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Benjamin Javillier, Principal Investigator, University of Liege
Other Study IDs: LPECarotide
Record Dates: First submitted 2019-11-19; First posted 2019-11-22 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Carotid Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LPEC/Sellick ultrasound
  Interventions: Procedure: Ultrasound LPEC/Sellick

INTERVENTIONS:
Procedure: Ultrasound LPEC/Sellick — We will perform an ultrasound of the carotid artery and then apply a Sellick manoeuvre and a left paratracheal compression of the cervical esophagus respectively.

SUMMARY:
Verify in ultrasound the impact of a Sellick and LPEC manoeuvre in terms of compression of the carotid artery and decrease in vascular flow.

ELIGIBILITY:
Inclusion Criteria:

* Adults Volunteers

Exclusion Criteria:

* pregnant women
* people with carotid artery defects
* people with an anomaly in the oropharyngeal massif

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Compression of the carotid artery during an esophageal compression manoeuvre | through study completion, an average of 1 month
  Measurement of the diameter of the carotid artery in cross-section and longitudinal section
Vascular flow of the carotid artery during an esophageal compression manoeuvre | through study completion, an average of 1 month
  Measurement of systolic velocities in pulsed Doppler in the carotid artery

SECONDARY OUTCOMES:
Measurement of the force to be applied to compress the esophagus without compressing the carotid artery | through study completion, an average of 1 month
  use of a dynamometer to measure the force required to exert at the left paratracheal level

CONTACTS AND LOCATIONS:
Locations (1):
- Javillier, Liège, Belgium